CLINICAL TRIAL: NCT07311876
Title: Clinical Lymphedema Evaluation - Advancing Reconstruction of Head and Neck Lymphatics With Symani
Acronym: CLEAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MMI (Medical Microinstruments, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-00148
Record Dates: First submitted 2025-12-23; First posted 2025-12-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lymphedema; Lymphedema of Face; Internal Lymphedema; External Lymphedema; Lymphedema of Neck
Keywords: lymphedema; head and neck lymphedema; symani
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Head and Neck Lymphedema (Experimental): The patients selected for the CLEAR Study will be adults over 22 years of age with a clinical indication for a microsurgical anastomosis of vessels between 0.1 and 2.5 mm in conjunction with lymphatic reconstruction of the head and neck.
  Interventions: Device: Symani Surgical System

INTERVENTIONS:
Device: Symani Surgical System — Symani® Surgical System is intended to perform surgical techniques during open microsurgical procedures.

SUMMARY:
The objective of this study is to evaluate the Symani System's safety and effectiveness for microsurgical anastomosis during open lymphatic reconstruction in the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. At least 22 years of age
2. Patients with acquired head and neck lymphedema with external lymphedema or both external and internal lymphedema
3. Patient agrees to participate in the study, return for all required follow-up visits, complete all study procedures, and has willingly provided written informed consent after receiving all information related to the study, its requirements, and the robotic-assisted procedure
4. Patient has a clinical indication for a microsurgical anastomosis of vessels between 0.1 and 2.5 mm in conjunction with lymphatic reconstruction of the head and neck
5. Patient has been compliant with complete decongestive therapy (CDT) for at least 4 weeks
6. Patient has undergone lymphatic mapping of the head and neck and functional lymphatic structures for reconstruction have been identified
7. Investigator deems the candidate acceptable for lymphatic reconstruction with a robotic-assisted microsurgical anastomosis in accordance with the Symani System's Instructions for Use (IFU)
8. Willingness to comply with recommended regimen of self-care, with consistent use of manual lymph drainage and/or appropriately sized compression garments from screening through the entire study duration (through the 6-month follow-up visit).

Exclusion Criteria:

1. Patient who is incapable and/or unwilling to provide informed consent
2. Patients with irreversible head and neck lymphedema, defined as stage 3 of the MD Anderson Cancer Center Head and Neck Lymphedema Rating Scale
3. Active systemic infection under treatment with intravenous antibiotics
4. Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders, previous mental disorders, or other disorders that may significantly affect the data collection or the ability to comply with the protocol per the investigator's discretion
5. Known history of significant bleeding, coagulopathy, or Von Willebrand's disease
6. Currently receiving chemotherapy or radiation therapy (uncontrolled tumor)
7. A history of malignancy or cancer treatment within the past 6 months (tumor control)
8. Patient with unsatisfactory manual lymphatic drainage and/or compression garments for at least six months
9. Patient with prior lymphatic reconstruction in the targeted head & neck area
10. Patient's lymphatic disease is due to lipedema
11. Patients with other medical conditions that could result in symptoms which overlap symptoms of lymphedema (e.g., thrombosis in the external or internal jugular vein)
12. Current infection in the head & neck area in which lymphedema is present
13. Currently enrolled in any other investigational clinical studies that the investigator believes may impact patient safety or outcomes
14. Patient is ineligible to participate for other reasons in the judgement of the investigator

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-03-28 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
Intraoperative anastomosis patency prior to closure. | The duration of the participants' index procedure.
  Intraoperative anastomosis patency prior to closure will be measured for each robotic anastomosis using indocyanine green (ICG) fluorescence imaging and will be evaluated prior to closure of the procedure site during the index procedure.
Freedom from device-related adverse events | The duration of the participants' index procedure through 30 days.
  All adverse events will be evaluated from the start of the index procedure through 30 days post index procedure.

SECONDARY OUTCOMES:
Change in flow pathways | From the pre-operative visit through 6 months post index procedure.
  Change in flow pathways will be assessed by an ICG lymphangiography
Change in MD Anderson Lymphedema Rating Scale for facial lymphedema | From the pre-operative visit through 6 months post index procedure.
  Scale ranges from 0-3, the higher score indicating worse disease state.
Assessment of Lymphedema of the Head and Neck Area (ALOHA) method for lymphedema measurement | From the pre-operative visit through 6 months post index procedure.
Change in Head and Neck Lymphedema and Fibrosis Symptom Inventory | From the pre-operative visit through 6 months post index procedure.
  It contains 33 items (symptoms) which are answered Yes or No. If the response is Yes to any given item, the patient is asked to rate the intensity of the symptom on a 5-point Likert scale. Each symptom then receives a score ranging from 0 (does not experience the symptom) to 5 (experiences the symptom with severe intensity).
Change in internal lymphedema | From the pre-operative visit through 6 months post index procedure.
  Assessed by Fiberoptic Endoscopic Evaluation of Swallowing (FEES) Examination
Technical Success | The duration of the participants' index procedure.
  as freedom from any device malfunction resulting in unplanned conventional (manual) suturing
All-cause readmission rates | The duration of the participants' index procedure through 30 days post index proceudre.
Procedure-related adverse events (AEs) rate | The duration of the participants' index procedure through 30 days post index proceudre.
Serious adverse events (AEs) rate | The duration of the participants' index procedure through 30 days post index proceudre.
Anastomosis-specific reoperation rate | The duration of the participants' index procedure through 30 days post index proceudre.